CLINICAL TRIAL: NCT04963725
Title: Symptom Improvement of Ulcerative Colitis After an Induction Dose of Ustekinumab in Japanese Clinical Practice, Measured Using Patient-Reported Outcomes
Brief Title: A Study of Symptom Improvement of Ulcerative Colitis After an Induction Dose of Ustekinumab in Japanese Clinical Practice
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108984; CNTO1275UCO4004 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-07-08; First posted 2021-07-15 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants Initiating Therapy with Ustekinumab: Data will be collected for participants in Japan who have had an inadequate response, or been intolerant to, conventional or biologic therapies. The treating physician has made the decision to initiate ustekinumab induction therapy in the routine clinical practice - either as a first or subsequent biologic therapy initiating for their moderate to severe ulcerative colitis.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — No intervention or treatment will be administered as part of this study. Data available per routine clinical practice at clinic visits as well as directly from participant using a smartphone/tablet application will be collected.

SUMMARY:
The purpose of this study is to describe the initial response to ustekinumab induction treatment for ulcerative colitis (UC) in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of ulcerative colitis (UC) in accordance with local practice
* Has a current UC severity that is judged by the treating physician to be moderate to severe (being a partial Mayo score of 5 to 9, inclusive)
* A decision has been made by the treating physician and the participant within routine clinical practice to commence treatment with ustekinumab, having been deemed to have an inadequate response to, or intolerant to, previous UC therapy
* Must sign an informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements. If the participant is 16 to 19, informed consent might be obtained from each study participant according to the regulation of institution/hospital and their legally acceptable representative must sign an ICF
* Must be able to read, understand, and complete participant-reported outcome instruments, and intend to cooperate with completion of participant-reported outcome instruments using smartphone/tablet

Exclusion Criteria:

* Has ever previously received ustekinumab (including clinical trial use)
* Are currently receiving, or have received within the past 3 months, systemic treatment with a biologic therapy for any other indication (example Crohn's disease, psoriasis, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis)
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 3 months before the start of the study or the first data collection time point
* Currently enrolled in an interventional study or another Janssen-sponsored observational study (including post-marketing surveillance)
* Based on physician judgement has i) severe extensive colitis and is at imminent risk of colectomy OR ii) a stoma or history of a fistula OR iii) previously had extensive colonic resection (example, less than 30 centimeter (cm) of colon remaining) OR iv) current fulminant colitis OR v) currently hospitalized for worsening of UC-related symptoms (not excluded if the reason for hospitalization is first dose of ustekinumab)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of participants who have had previously inadequate response, or have been intolerant to, conventional or biologic therapies and will be initiating ustekinumab for their ulcerative colitis.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-07-18 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With a Rectal Bleeding Score of 0 or 1 | Up to Week 8
  The rectal bleeding scores of 0 and 1 using physician's global assessment will be reported where 0 indicates 'No blood seen' and 1 indicates 'Streaks of blood with stool less than half the time'.
Percentage of Participants With a Stool Frequency Score of 0 or 1 | Up to Week 8
  The stool bleeding scores of 0 and 1 using physician's global assessment will be reported where 0 will indicate 'Normal number of stools' and 1 will indicate '1 to 2 stools more than normal'.

SECONDARY OUTCOMES:
Change From Baseline in Rectal Bleeding Score Through Week 8 | Baseline, Up to Week 8
  Change from baseline in rectal bleeding score through Week 8 will be reported.
Change from Baseline in Stool Frequency Score Through Week 8 | Baseline, Up to Week 8
  Change from baseline in stool frequency score through Week 8 will be reported.
Percentage of Participants with a Reduction in Rectal Bleeding Score of Greater than or Equal to (>=) 1 From Baseline | Up to Week 8
  Percentage of participants with a reduction in rectal bleeding score of >= 1 from baseline through Week 8 will be reported.
Percentage of Participants with Reduction in Stool Frequency Score of >= 1 From Baseline | Up to Week 8
  Percentage of participants with a reduction in stool frequency score of >= 1 from baseline through Week 8 will be reported.
Change from Baseline in Calculated Partial Mayo Score at Week 8 and Week 16 or Week 20 | Baseline, Week 8 and Week 16 or Week 20
  The partial Mayo (pMayo) is a composite score to indicate ulcerative colitis status without the requirement for endoscopy. It records participant-reported stool frequency over three days relative to normal on a 0-3 subscale (stool frequency, rectal bleeding, and physician global assessment of disease severity) each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores indicating more severe disease.
Change from Baseline in Rectal Bleeding Score at Week 16 or Week 20 | Baseline, Week 16 or Week 20
  Change from baseline in rectal bleeding score Week 16 or Week 20 will be reported.
Change from Baseline in Stool Frequency Score at Week 16 or Week 20 | Baseline, Week 16 or Week 20
  Change from baseline in stool frequency score at Week 16 or Week 20 will be reported.
Change from Baseline in Abdominal Pain Through Week 8 | Baseline, Up to Week 8
  Change from baseline in abdominal pain through Week 8 will be reported. Abdominal Pain will be evaluated based on numeric rating scale (NRS) ranging from 0 to 10 with lower score of 0 indicating 'no pain', score of 5 indicating 'moderate pain' and higher score of 10 indicating 'worst pain'. The abdominal pain score represents the most severe pain of the day.
Percentage of Participants with Presence of Nocturnal Diarrhea | Up to Week 8
  Percentage of participants with presence of nocturnal diarrhea will be reported. Nocturnal Diarrhea will be evaluated based on 'Yes/No' questionnaire, completed by participants using a smartphone/tablet-based application.
Percentage of Participants with Presence of Tenesmus | Up to Week 8
  Percentage of participants with presence of tenesmus will be reported. Tenesmus will be evaluated based on 'Yes/No' questionnaire, completed by participants using a smartphone/tablet-based application.
Percentage of Participants with Perceived Improvement in Ulcerative Colitis (UC) | Up to Week 8
  Percentage of participants with perceived improvement in UC will be reported. Perceived Improvement in UC will be evaluated based on NRS ranging from 0 to 10 with lower score of 0 indicating 'completely better (no UC symptoms)', score of 5 indicating 'starting condition (condition immediately before the induction of ustekinumab)' and higher score of 10 indicating 'poor condition (lots of UC symptoms).' Improvement is shown by recording a number less than 5 and worsening by recording a number greater than 5.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (23):
- Japan (23):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Juntendo University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Toho University Sakura Medical Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Hamamatsu University Hospital, Hamamatsu
  - Shimane University Hospital, Izumo
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Saitama Medical University Saitama Medical Center, Kawagoe
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Nagoya University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Ishida Clinic of IBD and Gastroenterology, Ōita
  - Shiga University of Medical Science Hospital, Ōtsu
  - Sapporo Medical University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Tokyo Yamate Medical Center, Shinjuku-ku
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Toyama Prefectural Central Hospital, Toyama
  - Yokkaichi Hazu Medical Center, Yokkaichi

REFERENCES:
- [Derived] Matsuoka K, Nagano K, Nagasaki S, Murata Y, Hisamatsu T. Symptom Improvement of ulceRative colitis after an Induction dose of UStekinumab in Japanese clinical practice (SIRIUS), measured using patient-reported outcomes: a prospective observational study. BMJ Open. 2022 May 4;12(5):e060081. doi: 10.1136/bmjopen-2021-060081. PMID 35508346